CLINICAL TRIAL: NCT00438659
Title: Phase III Randomized Double-Blind Study of Mometasone Furoate Versus Placebo in the Prevention of Radiation Dermatitis in Breast Cancer Patients Receiving Radiation Therapy
Brief Title: Mometasone Furoate in Preventing Radiation Dermatitis in Patients Undergoing Radiation Therapy to the Breast or Chest Wall for Invasive Breast Cancer or Ductal Carcinoma in Situ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Central Cancer Treatment Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Alliance for Clinical Trials in Oncology (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N06C4; NCI-2012-02708 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000530309 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Dermatologic Complications; Radiation Toxicity; Skin Reactions Secondary to Radiation Therapy
Keywords: dermatologic complications; skin reactions secondary to radiation therapy; radiation toxicity; breast cancer in situ; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer; ductal breast carcinoma in situ; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries; Breast Carcinoma In Situ; Breast Neoplasms, Male; Carcinoma, Intraductal, Noninfiltrating | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone (Experimental): Patients apply 2.5 mL mometasone furoate cream once daily to the treatment area (breast or chest wall) for the duration of planned radiotherapy.
  Interventions: Drug: mometasone furoate
- Placebo (Placebo Comparator): Patients apply 2.5 mL of an identical-appearing placebo cream to the treatment area as in arm I.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: mometasone furoate — Applied to treatment area
  Arms: Mometasone
Other: placebo — Applied to treatment area
  Arms: Placebo

SUMMARY:
RATIONALE: Steroid therapy, such as mometasone furoate, may prevent radiation dermatitis caused by radiation therapy. It is not yet known whether mometasone furoate is more effective than a placebo in preventing radiation dermatitis.

PURPOSE: This randomized phase III trial is studying mometasone furoate to see how well it works compared to a placebo in preventing radiation dermatitis in patients undergoing radiation therapy to the breast or chest wall for invasive breast cancer or ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of mometasone furoate vs placebo, in terms of decreased maximal severity of radiation dermatitis, in patients undergoing primary or adjuvant radiotherapy to the breast or chest wall for invasive breast cancer or ductal carcinoma in situ.

Secondary

* Compare the incidence of severe (grade ≥ 3) radiation dermatitis in patients treated with these drugs.
* Compare the time to onset and duration of severe radiation dermatitis in these patients.
* Assess skin toxicity and quality of life of these patients.
* Assess the adverse event profile of mometasone furoate in these patients.
* Compare skin toxicity data, in terms of provider-completed and patient-reported assessments, of patients treated with these drugs.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to radiation field (breast [post-lumpectomy] vs chest wall [post-mastectomy]), regional lymph nodes (treated vs not treated), and planned total radiation dose (including boost) (50-55 Gy vs > 55 Gy). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients apply mometasone furoate cream once daily to the treatment area (breast or chest wall) for the duration of planned radiotherapy.
* Arm II: Patients apply an identical-appearing placebo cream to the treatment area as in arm I.

Patients complete questionnaires and a symptom experience diary at baseline and periodically during study for quality of life, skin toxicity, and adverse event assessment.

After completion of radiotherapy, patients are followed for 2 weeks.

PROJECTED ACCRUAL: A total of 148 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of primary invasive breast cancer or ductal carcinoma in situ
* Planning to undergo ≥ 5 weeks of continuous definitive or adjuvant external-beam radiotherapy to 1 of the following sites:

  * Whole breast (as part of breast-conservation therapy)
  * Chest wall (as part of post-mastectomy irradiation)

    * Treatment of regional lymph nodes (i.e., axillary, supraclavicular, or internal mammary) allowed
* Must meet the following criteria for planned radiotherapy:

  * Planned total radiation dose ≥ 5,000 Gy and daily radiation dose between 1.75 and 2.12 Gy
  * No planned split-course radiotherapy
  * No partial breast treatment, defined as treatment of < 75% of the breast parenchyma
  * Intensity-modulated radiotherapy planning and delivery, conventional radiotherapy, or 3-dimensional radiotherapy techniques allowed
* Must be entered on study within 7 days prior to beginning radiotherapy

  * Must start study drug prior to receiving the third radiotherapy fraction
* No preexisting skin breakdown within the planned radiotherapy field at the time of study entry
* No bilateral breast cancer treatment
* No inflammatory carcinoma of the breast
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to complete questionnaires independently or with assistance
* No known allergy or hypersensitivity to mometasone furoate (Elocon® or generic cream), imidazolidinyl urea, or formaldehyde

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to the planned radiotherapy treatment area
* No concurrent or planned leukotriene inhibitors, including the following:

  * Zafirleukast
  * Monteleukast
  * Zileuton
* No concurrent or planned use of any prescription or over-the-counter medications containing hydrocortisone or any other cortisone or steroid-containing preparations (systemic, local, or topical) including, but not limited to, the following creams or ointments:

  * Cortaid®
  * Cortizone 10®
  * Tucks®
  * Preparation H®
* No other concurrent topical agents (e.g., lotions, aloe vera) to radiotherapy field during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Miller, MD, Study Chair — Mayo Clinic; Patricia Griffin, MD, Study Chair — Gibbs Regional Cancer Center at Spartanburg Regional Medical Center; James A. Martenson, MD, Study Chair — Mayo Clinic
Locations (189):
- United States (189):
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Background] Atherton PJ, Burger KN, Loprinzi CL, Neben Wittich MA, Miller RC, Jatoi A, Sloan JA. Using the Skindex-16 and Common Terminology Criteria for Adverse Events to assess rash symptoms: results of a pooled-analysis (N0993). Support Care Cancer. 2012 Aug;20(8):1729-35. doi: 10.1007/s00520-011-1266-x. Epub 2011 Sep 16. PMID 21922203
- [Result] Miller RC, Schwartz DJ, Sloan JA, Griffin PC, Deming RL, Anders JC, Stoffel TJ, Haselow RE, Schaefer PL, Bearden JD 3rd, Atherton PJ, Loprinzi CL, Martenson JA. Mometasone furoate effect on acute skin toxicity in breast cancer patients receiving radiotherapy: a phase III double-blind, randomized trial from the North Central Cancer Treatment Group N06C4. Int J Radiat Oncol Biol Phys. 2011 Apr 1;79(5):1460-6. doi: 10.1016/j.ijrobp.2010.01.031. Epub 2010 Aug 26. PMID 20800381
- [Result] Neben-Wittich MA, Atherton PJ, Schwartz DJ, Sloan JA, Griffin PC, Deming RL, Anders JC, Loprinzi CL, Burger KN, Martenson JA, Miller RC. Comparison of provider-assessed and patient-reported outcome measures of acute skin toxicity during a Phase III trial of mometasone cream versus placebo during breast radiotherapy: the North Central Cancer Treatment Group (N06C4). Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):397-402. doi: 10.1016/j.ijrobp.2010.05.065. Epub 2010 Oct 1. PMID 20888137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 176 patients were enrolled on this trial between 9/21/07 and 12/07/2007. There were 7 cancels (5 in Arm A and 2 in Arm B) and 3 patients discontinued treatment (1 in Arm A and 2 in Arm B). In total 84 in Arm A and 82 in Arm B were evaluable for the primary endpoint.
Groups:
- Placebo: Patients apply 2.5 mL of an identical-appearing placebo cream to the treatment area as in arm A.
Period: Overall Study
Arm/Group | Mometasone | Placebo
Started | 90 | 86
Completed | 84 | 82
Not Completed | 6 | 4
Not completed — Discontinued Mometasone/Placebo | 1 | 2
Not completed — Cancel | 5 | 2

BASELINE CHARACTERISTICS:
Population: All (169) eligible patients are included in the baseline analysis. There were 5 cancels in Arm I and 2 in Arm II.
Groups:
- Placebo: Patients apply 2.5 mL of an identical-appearing placebo cream to the treatment area as in arm B.
- Total: Total of all reporting groups
Arm/Group | Mometasone | Placebo | Total
Number analyzed (Participants) | 85 | 84 | 169
Age, Continuous [Median (Full Range); unit: years] | 60 (14.63) [35 to 89] | 57 (11.8) [27 to 85] | 59 (13.29) [27 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 84 | 169
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 85 | 84 | 169

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Grade of Radiation Dermatitis by Treatment Arm.
Description: Maximum grade of radiation dermatitis as measured by the Common Terminology Criteria (CTCAE) for Adverse Events (AE), Version 3.0. Grade 1 (Mild AE), Grade 2 (Moderate AE), Grade 3 (Severe AE), Grade 4 (Life-threatening or disabling AE), Grade 5 (Death related to AE).
Time Frame: During Radiation Treatment, up to a maximum of 9 weeks.
Measure: Mean (Full Range); unit: Grade
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 84 | 82
Grade | 1.2 [0.0 to 3.0] | 1.3 [0.0 to 3.0]
Statistical Analysis 1: Comparison: Mometasone vs Placebo; Test type: Superiority or Other; p = 0.18, t-test, 2 sided

2. Secondary Outcome: Incidence of Severe ( Grade >=3) Radiation Dermatitis
Description: To compare incidence of severe (Grade ≥ 3) radiation dermatitis as measured by the CTCAE v3.0 for the mometasone and placebo arms.
Time Frame: During Radiation Treatment, up to a maximum of 9 weeks.
Measure: Number; unit: Paticipants
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 84 | 82
Paticipants
  Did not experience grade >=3 radiation dermatitis | 80 | 78
  Experience grade >=3 radiation dermatitis | 4 | 4

3. Secondary Outcome: Skin Toxicity as Measured by the Skin Toxicity Assessment Tool
Description: Mean of the Maximum Patient Reported Skin Toxicity Assessment Tool (STAT) per patient on a 0 to 5 scale during radiation treatment. Lower scores indicate less toxicity.
Time Frame: During Radiation Treatment, up to a maximum of 9 weeks.
Measure: Mean (Standard Deviation); unit: Score on a 0 to 5 scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 83 | 84
Score on a 0 to 5 scale
  STAT: Discomfort/Burning | 1.5 (1.69) | 2.1 (1.74)
  STAT: Itching | 1.5 (1.53) | 2.2 (1.47)
  STAT: Pulling | 1.0 (1.36) | 1.4 (1.66)
  STAT: Discomfort/Tenderness | 2.1 (1.57) | 2.5 (1.61)

4. Secondary Outcome: Skin Toxicity as Measured by a Dermatologic Quality-of-life Instrument (Skindex-16).
Description: Patient-Reported Mean of the Maximum Total a Skindex-16 Toxicity Score per patient on a 0-6 scale during radiation treatment (Lower score indicates less toxicity).
Time Frame: During Radiation Treatment, up to a maximum of 11 weeks.
Measure: Mean (Standard Deviation); unit: score on a 0-6 scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 83 | 84
score on a 0-6 scale | 1.4 (1.24) | 1.7 (1.35)

5. Secondary Outcome: Duration of Severe (Grade ≥ 3) Radiation Dermatitis as Measured by the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. This Analysis Was Not Completed Due to Too Little Incidence of the Dermatitis.
Description: To compare time to onset and duration of severe (Grade ≥ 3) radiation dermatitis as measured by the CTCAE v3.0 for the mometasone and placebo arms. This analysis was not completed due to too little incidence of the dermatitis.
Time Frame: During Radiation Treatment, up to a maximum of 9 weeks.
Population: This analysis was not completed due to too little incidence of the dermatitis.
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Quality of Life (QOL) as Measured by Linear Analogue Self-Assessment (LASA)
Description: Patient completed QOL assessment was the Linear Analogue Self-Assessment (LASA). This instrument consisted of 6 questions with responses ranging from 0 (poor QOL) to 100 (best QOL).
Time Frame: During Radiation Treatment, up to a maximum of 11 weeks.
Population: Patients who completed at least 1 assessment were evaluable for this secondary end point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 85 | 84
units on a scale | 85 (16) | 82 (19)

7. Secondary Outcome: QOL Domains as Measured by LASA
Description: Mean scores of Linear Analogue Sef-Assessment (LASA) Mental, physical, emotional, social, spiritual wel-being on a 0 (as bad as it can be) to 100 (as good as it can be) scale.
Time Frame: During Radiation Treatment, up to a maximum of 11 weeks.
Population: Patients who completed at least 1 assessment were evaluable for this secondary end point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 85 | 84
units on a scale
  Mental well-being | 86 (15) | 84 (18)
  Physical well-being | 83 (17) | 79 (19)
  Emotional well-being | 85 (16) | 80 (19)
  Social well-being | 81 (19) | 77 (24)
  Spiritual well-being | 89 (14) | 84 (21)

8. Secondary Outcome: Adverse Events Assessed Clinically by NCI CTCAE v3.0
Time Frame: During Radiation Treatment, up to a maximum of 9 weeks.
Measure: Number; unit: participants
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 84 | 82
participants
  ARTHRALGIA: Severe | 1 | 0
  BURN: Mild | 32 | 32
  BURN: Moderate | 6 | 5
  BURN: Severe | 0 | 2
  CELLULITES INFECTN: Moderate | 1 | 1
  COUGH: Severe | 0 | 1
  DERMATOLOGY: Mild | 11 | 19
  DERMATOLOGY: Moderate | 8 | 3
  DERMATOLOGY: Severe | 0 | 2
  FATIGUE: Moderate | 0 | 1
  PAIN: Severe | 0 | 1
  PAIN-BREAST: Moderate | 1 | 1
  PAIN-CHEST: Moderate | 0 | 1
  PRURITUS: Mild | 36 | 50
  PRURITUS: Moderate | 14 | 14
  PRURITUS: Severe | 1 | 5
  SKIN ATROPHY: Mild | 0 | 2
  SKIN ATROPHY: Moderate | 1 | 0
  SKIN HYPOPIGMENT: Mild | 5 | 8
  SKIN HYPOPIGMENT: Moderate | 1 | 1
  SKIN IRRITATION: Moderate | 0 | 1
  SKIN STRIAE: Mild | 2 | 6
  SKIN STRIAE: Moderate | 1 | 0

9. Secondary Outcome: Adverse Events Reported by the Patient in the Symptom Experience Diary (SED).
Description: Maximum SED score during radiation treatment per patient on a 0 to 10 scale (lower score is better)
Time Frame: During Radiation Treatment, up to a maximum of 11 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mometasone | Placebo
Number analyzed (Participants) | 83 | 84
units on a scale
  Redness | 5.1 (3.52) | 6.8 (3.34)
  Dry Peeling | 2.7 (3.33) | 3.1 (3.66)
  Wet Peeling | 1.3 (2.65) | 1.6 (3.14)
  Weeping | 1.2 (2.77) | 1.4 (2.86)
  Rash | 2.6 (3.38) | 4.0 (3.96)
  Swelling | 2.3 (3.29) | 2.4 (3.14)
  Fatigue | 4.5 (3.06) | 5.0 (3.11)
  Decrease in color | 2.3 (3.12) | 2.1 (2.81)
  Band, Stripes or Lines | 1.7 (2.8) | 1.5 (2.66)

ADVERSE EVENTS:
Arm/Group | Mometasone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/82
Other Adverse Events (participants affected / at risk) | 75/84 | 81/82
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone (N=84) | Placebo (N=82)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 64 (235) | 69 (263)
Thermal burn (Injury, poisoning and procedural complications) | 38 (83) | 39 (81)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Atrophy skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 51 (137) | 69 (214)
Skin disorder (Skin and subcutaneous tissue disorders) | 19 (42) | 25 (48)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 6 (14) | 9 (21)
Skin striae (Skin and subcutaneous tissue disorders) | 3 (12) | 6 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes